CLINICAL TRIAL: NCT02942615
Title: A Randomized Multi-center Phase III Study About the Safety Management of Cardiac Toxicity in Breast Cancer Patients Under Multidiscipline Therapy.
Brief Title: The Safety Management of Cardiac Toxicity in Breast Cancer Patients Under Multidiscipline Therapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 6th People's Hospital (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Jiayi Chen, Chief of department of radiation oncology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Cardio-RT
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Breast Neoplasms; Cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart safety management (Experimental): limit heart dose more frequent follow up of cardiac function professional management of cardiac toxicity
  Interventions: Other: limit heart dose
- Control group (No Intervention): without any restrict heart dose limitation for RT Follow up of cardiac function Observation and without any special management of cardiac toxicity

INTERVENTIONS:
Other: limit heart dose — limit heart dose: Dmean≤6Gy,V30≤20%,V10≤50%
  Other Names: frequently follow of cardiac function; management of cardiotoxicity
  Arms: Heart safety management

SUMMARY:
This trial is to explore the optimal strategies for guaranteeing the cardiac safety of breast cancer patients following adjuvant radiotherapy in the modern era of multidisciplinary treatment.

DETAILED DESCRIPTION:
With the development of modern radiotherapy techniques, the dose-volume of heart irradiated could be kept in much low level. However, until now, the optimal dose-volume parameters for limiting heart irradiation, the optimal follow-up interval for cardiac safety after adjuvant radiotherapy, the optimal screening examinations and treatments for irradiation-induced cardiac toxicity are unclear. We designed this trial to find answer for above questions to establish rationalization proposal for prevention, treatment and follow-up for cardiac toxicity associated with adjuvant radiotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate the research and sign the informed consent file;
* Patients aged 18-80 years;
* KPS≥70;
* Pathological diagnosis for invasive breast cancer;
* Patients received anthracycline/paclitaxel based chemotherapy, or herceptin based targeted therapy;
* No functional heart disease;
* LVEF≥50%;
* Patients received breast conserving surgery;
* Patients received modified radical mastectomy: T1-2 with N1-3 or T3-4 with any N;
* Tumor margin negative;
* No metastases;
* No other malignant tumor history.

Exclusion Criteria:

* Patients with metastases;
* Tumor margin positive;
* Patients received modified radical mastectomy with T1-2 and N0;
* Patients have other malignant tumor;
* Patients have a history of heart disease;
* Patients received chest radiotherapy previously;
* Patients with severe organic and functional disease;
* Unqualified patients with sufficient reasons;
* Cannot or no willing to sign the informed consent file;
* Patients with autoimmune disease;
* Women with pregnancy, planned pregnancy or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
cardiac toxicity event free survival | 1 year
  The time from the date of randomization to any recurrence of clinical or subclinical cardiac toxicity

SECONDARY OUTCOMES:
cardiac toxicity event free survival | 5 years
  The time from the date of randomization to any recurrence of clinical or subclinical cardiac toxicity
cardiac toxicity event free survival | 10 years
  The time from the date of randomization to any recurrence of clinical or subclinical cardiac toxicity
overall survival | 5 years
  The time from the date of randomization to the date of death from any cause
overall survival | 10 years
  The time from the date of randomization to the date of death from any cause
relative change of value of serum cardiac biomarkers of creatine kinase (CK)-MB | 1 year
  The change of value of serum cardiac biomarkers during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of value of serum cardiac biomarkers of Cardiac troponin (cTn)-I | 1 year
  The change of value of serum cardiac biomarkers during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of value of serum cardiac biomarkers of N-terminal pro brain natriuretic peptide (NT-proBNP) | 1 year
  The change of value of serum cardiac biomarkers during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of value of serum cardiac biomarkers of CK-MB | 5 years
  The change of value of serum cardiac biomarkers during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of value of serum cardiac biomarkers of cTn-I | 5 years
  The change of value of serum cardiac biomarkers during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of value of serum cardiac biomarkers of NT-proBNP | 5 years
  The change of value of serum cardiac biomarkers during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of left ventricular ejection fraction (LVEF) | 1 year
  The change of value of LVEF during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of LVEF | 5 year
  The change of value of LVEF during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapyThe change of value of LVEF during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
relative change of LVEF | 10 year
  The change of value of LVEF during and after adjuvant radiotherapy compared with baseline before initiation of adjuvant radiotherapy
Quality of Life-EORTC QLQ-C30 | 1 year
  Quality of life will be assessed using self-administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC QLQ-BR23 | 1 year
  Quality of life will be assessed using self-administered questionnaire EORTC QLQ-BR23
Quality of Life-EORTC QLQ-C30 | 5 years
  Quality of life will be assessed using self-administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC QLQ-BR23 | 5 years
  Quality of life will be assessed using self-administered questionnaire EORTC QLQ-BR23

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China